CLINICAL TRIAL: NCT00918229
Title: One-arm, Multi-center, International Prospective Study to Assess the Safety and Efficacy of BioProtect Biodegradable Implantable Balloon in Prostate Cancer Subjects Undergoing Radiotherapy
Brief Title: Pilot Study to Assess the Safety and Efficacy of BioProtect Balloon in Prostate Cancer Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BPI-01 (USA)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Prostate; cancer; radiation; biodegradable implantable balloon; intrarectal balloon
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- balloon implantation (Other): implantation of an absorbable perirectal spacer balloon
  Interventions: Device: balloon implant; Procedure: Balloon implantation

INTERVENTIONS:
Device: balloon implant — Absorbable perirectal spacer implantation
Procedure: Balloon implantation — Implantation of the balloon between the prostate and the anterior rectal wall

SUMMARY:
Primary Goal

The study's primary goal is to assess the safety of the BioProtect biodegradable balloon implant and implantation procedure, in prostate cancer subjects undergoing routine radiation therapy (XRT) treatment. Safety of the BioProtect device will be assessed by reporting adverse events.

Secondary Goal

The study's secondary goal is to evaluate the effectiveness of the BioProtect biodegradable balloon implant in prostate cancer subjects undergoing routine XRT treatment. Effectiveness will be assessed in terms of increased distance between anterior rectal wall and prostate and noticeable reduction of isodose to the rectum.

DETAILED DESCRIPTION:
Primary Endpoint Parameters

The incidence of unexpected serious adverse events related to BioProtect's SpaceGuard balloon implant and/or implantation procedure:

1. Serious Adverse Events related to the BioProtect balloon and/or implantation procedure were defined by the Clinical Trials.gov definition of a serious adverse event. Serious Adverse Events will be documented in Serious Adverse Event Form.
2. Adverse Events related to the BioProtect balloon and/or implantation procedure. Adverse Events were documented in Adverse Event Form.
3. Subjective discomfort related to the balloon and implantation procedure were assessed by a pain analogue scale.

Secondary Endpoint Parameters A 10% decrease or greater of the average rectal doses at V50 in at least 75% of the subjects after balloon implantation as compared to the doses at V50 before the balloon implantation. This was measured by routine Dose Volume Histogram (DVH) per local hospital practice and according to the instructions regarding anatomical landmarks delineated in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult male above 45 years old and less than 85.
* Diagnosed locally confined prostate cancer per hospital practice and definitions for local confined prostate cancer.
* Subject is scheduled for only localized prostate XRT treatments
* Zubrod performance status 0-1; or Karnofsy >80
* Blood CBC and biochemistry up to two weeks before screening demonstrating:

  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 10.0 g/dl
  * Normal values of electrolytes (sodium, potassium, calcium)
  * Normal values of the PT, PTT and INR tests.
* Peak Uroflow rate ≥ 13ml/sec
* Residual Urine volume Test result < 150 ml
* Urinalysis (RBC, WBC) and urine culture
* Subject able to comprehend and give informed consent for participation in this study and are considered by the investigator to have good compliance for the study.

Exclusion Criteria:

* Any prior prostate resection with a compliant prostate urethra as assessed by transrectal ultrasound (TRUS)
* Prior radical prostatectomy
* Prior cryosurgery or radiotherapy for prostate cancer, or other local therapy for prostate cancer
* Suspected extension of the prostate tumour toward the rectum as evidenced by acceptable imaging modalities used in the study site
* Prior surgical procedure involving peri-rectal and peri-prostatic area
* Prior radiotherapy to the pelvis, including brachytherapy at the same body organ
* Unstable angina
* Congestive heart failure (CHF) phase III or IV or CHF requiring hospitalization within the last 6 months prior to screening
* Transmural myocardial (MI) infarction within the last 6 months prior to screening
* Moderate to severe respiratory failure, hepatic failure or renal failure
* Acute infection requiring intravenous antibiotics at the time of screening
* Uncontrolled bleeding disorders
* Uncontrolled diabetes mellitus
* Known to be HIV positive or have any other immunosuppressive disorder
* Inflammatory diseases of the perineal skin
* Urinary tract infection or acute or chronic prostatitis
* Uncontrolled moderate to severe urinary disorders
* Active inflammatory bowel disease or moderate to severe gastrointestinal (GI) disorders
* Known or suspected rectal carcinoma
* Subjects after anterior resection of rectum or after rectal amputation
* Concurrent participation in any other clinical study

Intra-operative exclusion criteria:

* Irregular findings by the implanting physician before or during implantation that to the best of the implanting physician may lead to prostate compliance leading to urinary retention or other such symptoms.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Muncher, Dr., Study Director — BioProtect
Locations (1):
- Virginia Commonwealth University School of Medicine, Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Implantation: One arm study only
  implantation of an absorbable perirectal spacer balloon
  balloon implant: Absorbable perirectal spacer implantation
  Balloon implantation: Implantation of the balloon between the prostate and the anterior rectal wall
Period: Overall Study
Arm/Group | Balloon Implantation
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Implantation
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a Reduction of at Least 25% of the Volume of the Rectum Receiving at Least 70 Gy.
Description: Evaluated in subjects with prostate cancer who underwent radiotherapy by means of IMRT and who received the ProSpace, with individual patient success defined as a reduction of at least 25% of the volume of the rectum receiving greater or equal to 70 Gy (VRectum70) when compared to pre-implantation values.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Implantation
Number analyzed (Participants) | 24
Participants | 24

2. Secondary Outcome: Rate of Occurrence of Grade 2 or Greater Rectal Adverse Event or Procedure Related Adverse Events.
Description: Compare the rate of occurrence of rectal adverse events and implantation procedure related adverse events in balloon and control groups.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Implantation
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definition used did not differ from the clintrials.gov definition. All data was reviewed for the occurrence of these events. No serious events occurred.
Arm/Group | Balloon Implantation
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Implantation (N=24)
Bleeding (Renal and urinary disorders) | 1 (1) — Trace of blood in semen
Urinary retention (Renal and urinary disorders) | 1 (1) — Transient acute urinary retention, resolved in a few hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No